CLINICAL TRIAL: NCT02458183
Title: A Multinational, Multicenter, Randomized, Comparative, Open-label, Phase 3 Study to Assess the Immunogenicity and Safety of DTaP-IPV (Diphtheria-tetanus-acellular Pertussis-inactivated Poliovirus) Vaccine Administered to Healthy Infants
Brief Title: Vaccine -diphthEria -tetaNus -Acellular pertUssis-inactivated polioviruS
Acronym: Venus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BR-DTPP-CT-301
Record Dates: First submitted 2015-04-27; First posted 2015-06-01 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Diphtheria; Tetanus; Pertussis; Poliomyelitis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DTaP-IPV combination vaccine (Experimental): Dosage and administration: A 0.5-mL dose is administered intramuscularly in the anterol-ateral aspect of right thigh at the age of 2, 4, and 6 months
  Interventions: Biological: DTaP-IPV combination vaccine
- DTaP vaccine and IPV vaccine (Active Comparator): Product name: : Boryung DTaP Vaccine Inj. (Prefilled syringe) (Absorbed diphtheria, tetanus toxoid, and purified pertussis combination vaccine) Dosage and administration: A 0.5-mL dose is administered 3 times intramuscularly in the anterolateral aspect of right thigh at the age of 2, 4, and 6 months.
  Product name: IPVAX INJ. PREFILLED SYRINGE INJ. Dosage and administration: A 0.5-mL dose is administered intramuscularly in the anterol-ateral aspect of left thigh at the age of 2, 4, and 6 months.
  Interventions: Biological: DTaP vaccine and IPV vaccine

INTERVENTIONS:
Biological: DTaP-IPV combination vaccine — 0.5-mL IM
  Arms: DTaP-IPV combination vaccine
Biological: DTaP vaccine and IPV vaccine — 0.5-mL IM
  Other Names: Boryung DTaP Vaccine Inj. (Prefilled syringe); IPVAX INJ. PREFILLED SYRINGE INJ
  Arms: DTaP vaccine and IPV vaccine

SUMMARY:
The objective of this study is to assess the immunogenicity and safety of the DTaP-IPV combination vaccine compared with those of separate DTaP and IPV vaccines administered to healthy infants at 2, 4, and 6 months of age.

DETAILED DESCRIPTION:
A multinational, multicenter, randomized, comparative, open-label, phase 3 study

Primary Objective: To assess the vaccine response rates after the three-dose primary vaccination Secondary Objectives: To measure the antibody titer after the three-dose primary vaccination and to assess the safety of the investigational products

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian (legally authorized representative) has given voluntary written consent to the subject's participation after being fully informed of the purpose, methods, risks, and benefits of the study.
* Male and female infants reaching at least 7 weeks of age on the day of first dose of investigational product.
* Male and female infants who are identified to be healthy based on physical examination and medical history.

Exclusion Criteria:

* Subjects who have acute febrile illness with tympanic temperature of ≥38.0 ℃ on the day of vaccination.
* Subjects who have moderate or severe acute disease (regardless of fever).
* Subjects who have any history of diphtheria, tetanus, pertussis, or poliomyelitis.
* Subjects who have major congenital defects.
* Subjects who show any evidence of continuous hematologic, hepatic, cardiac, re-nal, or respiratory disease.
* Subjects who have abnormalities in the immune system, or congenital/acquired immune deﬁciency.
* Subjects who received immunosuppressive dose of systemic corticosteroids thera-py within 30 days before the vaccination.
* Subjects who are likely to have adverse side effects on central nervous system be-cause of the subjects' family history of genetic diseases in central nervous system such as progressive neurological problems or epilepsy.
* Subjects who are allergic to the ingredients of the investigational products.
* Subjects who have received immunoglobulins or blood products or plan to get those medications.
* Subjects who have received vaccines other than those allowed in the protocol or plan to get those prohibited vaccines during the study period.
* Subjects who are currently participating or planning to participate in other clinical studies during the study period.
* Other ineligible conditions judged at the discretion of principal investigators or subinvestigators.

Ages: 7 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 476 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Vaccine response rate | 4 weeks after the three-dose primary vaccination
  Vaccine response rate of anti-diphtheria, anti-tetanus, anti-PT, anti-FHA, and anti-poliovirus type 1, 2, 3 at 4 weeks after the completion of the final vaccination
  Criteria of vaccine response rate Anti-diphtheria: Antibody titer after the completion of the final vaccination ≥ 0.1 IU/mL anti-tetanus: Antibody titer after the completion of the final vaccination ≥ 0.1 IU/mL anti-PT, anti-FHA: Antibody titer at 4 weeks after the completion of the final vaccination is at least 4 times the baseline antibody titer anti-poliovirus type 1, 2, 3: Serum neutralizing antibody dilution ratio after the completion of the final vaccination ≥ 1:8

SECONDARY OUTCOMES:
Geometric mean titer (GMT) | 4 weeks after the three-dose primary vaccination
  anti-diphtheria, anti-tetanus, anti-PT, anti-FHA, and anti-poliovirus type 1, 2, 3 at 4 weeks after the completion of the final vaccination

OTHER OUTCOMES:
Solicited adverse event/adverse drug reaction | 24~26 weeks after the final vaccination
  Incidence of Treatment-Emergent Adverse Events
Unsolicited adverse event/adverse drug reaction | 24~26 weeks after the final vaccination
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: HJ Jung, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (20):
- South Korea (18):
  - Inje University Busan Paik Hospital, Busan
  - KeiMyung University Dongsan Medical Center, Daegu
  - Gwangmyeong Sungae Hospital, Gyeonggi-do
  - Wonkwang University Hospital, Iksan
  - Inha University Hospital, Incheon
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Cheil General Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Eulgi General Hospital, Seoul
  - Gangnam Sevrance Christian Hospital, Seoul
  - Hallym University Medical Center, Seoul
  - KEPCO Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - KyungHee University Hospital at Gangdong, Seoul
  - KyungHee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Wonju Sevrance Christian Hospital, Wŏnju
- Thailand (2):
  - Siriraj Hospital, Bangkok
  - Thammasat University, Bangkok

IPD SHARING:
Plan to Share IPD: No